CLINICAL TRIAL: NCT06939608
Title: Kinetics of Yohimbine in Humans to Explore Sex and CYP2D6 Genotype Interactions - YOKI-1 Study
Brief Title: Kinetics of Yohimbine in Humans to Explore Sex and CYP2D6 Genotype Interactions
Acronym: YOKI-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Stefan Engeli, MD, Prof. Dr. med Stefan Engeli, University Medicine Greifswald
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IPHA-2025-011
Record Dates: First submitted 2025-03-31; First posted 2025-04-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pharmacokinetic Study in Healthy Volunteers
Keywords: sex-specific differences; pharmacokinetics; yohimbine; CYP2D6; genetic polymorphisms; drug metabolism; CYP1A2; ¹³C₃-caffeine
MeSH Terms: interventions — Yohimbine; CID-1 proterin, C elegans

STUDY DESIGN:
Intervention Model Description: The study is designed as an open-label, four-arm, parallel assignment, single oral dose protocol, stratifying participants by CYP2D6 genotype (extensive vs. poor metabolizers) and biological sex (women vs. men).
Masking Description: This is an open-label study; no parties involved are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Women, Poor Metabolizers (PM) (Active Comparator): Participants in this arm are women, as identified by their sex assigned at birth, classified as poor metabolizers (PM) based on their CYP2D6 genotype. Poor metabolizers are homozygous for CYP2D6 *3, *4, *5, *6 or carry heterozygous combinations of these alleles. Participants were selected to achieve best matching between arms according to age, BMI, alcohol consumption and smoking.
  Interventions: Dietary Supplement: Yohimbine; Other: ¹³C₃-caffeine
- Women, Extensive Metabolizers (EM) (Active Comparator): Participants in this arm are women, as identified by their sex assigned at birth, classified as extensive metabolizers (EM) based on their CYP2D6 genotype. Extensive metabolizers are homozygous for CYP2D6 *1, *2, *35 or carry heterozygous combinations of these alleles. Participants were selected to achieve best matching between arms according to age, BMI, alcohol consumption and smoking.
  Interventions: Dietary Supplement: Yohimbine; Other: ¹³C₃-caffeine
- Men, Poor Metabolizers (PM) (Active Comparator): Participants in this arm are men, as identified by their sex assigned at birth, classified as poor metabolizers (PM) based on their CYP2D6 genotype. Poor metabolizers are homozygous for CYP2D6 *3, *4, *5, *6 or carry heterozygous combinations of these alleles. Participants were selected to achieve best matching between arms according to age, BMI, alcohol consumption and smoking.
  Interventions: Dietary Supplement: Yohimbine; Other: ¹³C₃-caffeine
- Men, Extensive Metabolizers (EM) (Active Comparator): Participants in this arm are men, as identified by their sex assigned at birth, classified as extensive metabolizers (EM) based on their CYP2D6 genotype. Extensive metabolizers are homozygous for CYP2D6 *1, *2, *35 or carry heterozygous combinations of these alleles. Participants were selected to achieve best matching between arms according to age, BMI, alcohol consumption and smoking.
  Interventions: Dietary Supplement: Yohimbine; Other: ¹³C₃-caffeine

INTERVENTIONS:
Dietary Supplement: Yohimbine — A single oral dose of 50 µg yohimbine, administered as 2 x 1 tablets of Yohimbinum hydrochloricum D4® will be co-administered with 25 mg of ¹³C₃-caffeine as drinking solution with 240mL of still water under overnight fasting conditions. A total of 19 blood samples will be collected at defined time points (baseline; 10; 20; 30; 40; 50; 60; 70; 80; 90; 100; 110 min; 2; 3; 4; 6; 8; 10; 24 h). At each time point, 4.9 mL of blood will be drawn for plasma separation to determine yohimbine, the primary metabolite 11-OH-yohimbine and ¹³C₃-caffeine with associated CYP1A2 dependent metabolites.
Other: ¹³C₃-caffeine — A single oral dose of 25 mg of ¹³C₃-caffeine as a drinking solution will be co-administered with yohimbine with 240 mL of still water under overnight fasting conditions. ¹³C₃-caffeine is a stable isotope-labeled standard probe for phenotyping CYP1A2 activity and assessing potential interactions between CYP2D6 and CYP1A2. Plasma concentrations of ¹³C₃-caffeine with associated CYP1A2 dependent metabolites will be measured at predefined time points, following the sampling schedule outlined for yohimbine.

SUMMARY:
This study investigates the pharmacokinetics of yohimbine in women and men aged 18 to 40 years to explore sex-specific differences in CYP2D6-dependent drug metabolism. Participants will be classified by their CYP2D6 genotype into extensive metabolizers (EM) and poor metabolizers (PM), forming four distinct study arms:

Arm 1) Women, Poor Metabolizers (PM) n=13 Arm 2) Women, Extensive Metabolizers (EM) n=5 Arm 3) Men, Poor Metabolizers (PM) n=13 Arm 4) Men, Extensive Metabolizers (EM) n=5

Each study arm will receive a single oral dose of 50 µg yohimbine (2 x 1 tablets, 25 µg per tablet) and 25 mg of ¹³C₃-caffeine co-administered as a drinking solution.

The purpose of this study is:

1. To characterize the pharmacokinetics of yohimbine following a single oral dose in women and men across different CYP2D6 phenotypes.
2. To evaluate yohimbine's suitability as a reliable probe for assessing CYP2D6 activity.
3. To investigate potential interactions between CYP2D6 and CYP1A2, as well as interindividual variability in CYP1A2-dependent caffeine metabolism.

DETAILED DESCRIPTION:
The study is designed as an open-label, single-dose protocol with four study arms based on sex and CYP2D6 genotype. A single oral dose of yohimbine and ¹³C₃-caffeine will be administered with 240 ml of still water under overnight fasting conditions.

A total of 19 blood samples will be collected at defined time points (baseline; 10; 20; 30; 40; 50; 60; 70; 80; 90; 100; 110 min; 2; 3; 4; 6; 8; 10; 24 h). At each time point, 4.9 mL of blood will be drawn for plasma separation to determine yohimbine, the primary metabolite 11-OH-yohimbine and 13C₃-caffeine with associated CYP1A2 dependent metabolites. One additional blood sample (EDTA tube) for potential future genetic analysis, will be collected together with the baseline kinetic samples.

For each participant, a total of approximately 98 mL of blood will be collected during the kinetic visits and an additional 12 mL during the screening visit.

Following the administration of yohimbine and 13C3-caffeine, participants will consume 200 mL of sparkling water every hour to stimulate gastrointestinal peristalsis facilitate substance transport. Two hours post-administration, participants may have a cup of tea or coffee, while a standardized meal will be served four hours after dosing.

Urine samples will be collected over 24 hours in three intervals (0-4 h, 5-10 h, 11-24 h). Blood pressure and heart rate monitoring will be conducted during the initial four hours and participants will remain in the Clinical Research Unit of the Institute of Pharmacology for the first 10 hours post-administration. At 24 hours post-dosing, participants will return to the Clinical Research Unit for the final scheduled blood collection and to provide their last urine sample (11-24 h).

ELIGIBILITY:
Inclusion Criteria:

1. individuals of both biological sexes, assigned as women or men at birth
2. age: ≥ 18 and ≤ 40 years
3. possesses the ability to understand the study purpose and design
4. contractually capable and provides signed informed consent form
5. in good general health or with mild and/or well-managed conditions such as allergies, asthma, hypertension or orthopedic diseases
6. taking no more than three chronic medications
7. individuals classified as either extensive metabolizers (EM) or poor metabolizers (PM) based on their CYP2D6 genotype:

Extensive Metabolizers (EM):

homozygous for CYP2D6 *1,CYP2D6 *2, CYP2D6 *35, or heterozygous combination of any of these alleles

Poor Metabolizers (PM):

homozygous for CYP2D6 *3, CYP2D6 *4, CYP2D6 *5, CYP2D6 *6, or heterozygous combination of any of these alleles

Exclusion Criteria:

1. BMI > 30 kg/m2 and < 18 kg/m2
2. body weight < 48 kg
3. women: known pregnancy or lactation period; positive urine pregnancy test at screening or kinetic visit
4. men: hemoglobin < 13 g/dl (8,07 mmol/l) women: hemoglobin < 12 g/dl (7,45 mmol/l)
5. elevated liver function tests (1 or more of ALAT, ASAT, yGT, Bilirubin > 2x ULN)
6. reduced renal function (eGFRMDRD < 60 mL/min/1,7 m2)
7. QTcF > 450 ms in screening ECG
8. current or recent psychiatric disorders requiring treatment including depression, bipolar disorder, schizophrenia, psychosis or severe anxiety disorders
9. drug dependency at the time of visit
10. use of recreational drugs more than twice a week
11. any known hypersensitivity or allergic reactions to yohimbine or caffeine
12. history of severe hypersensitivity reactions and/or anaphylaxis
13. poor venous conditions that make it impossible to place a peripheral venous catheter and regularly draw blood through it

o) intake of drugs interfering with CYP2D6 and/or CYP1A2 during the past seven days p) intake of yohimbine within 48 hours and caffeine within 16 hours prior to study participation q) engagement in extreme physical activity within 48 hours prior to study participation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Yohimbine plasma concentration expressed as area under the curve (AUC₀-₂₄h) - arm 1 vs. arm 3 | 24 hours
  Difference in plasma concentrations of yohimbine expressed as area under the curve (AUC₀-₂₄h) between women classified as CYP2D6 poor metabolizers (PM) (arm 1) and men classified as CYP2D6 poor metabolizers (PM) (arm 3).
Yohimbine plasma concentration expressed as area under the curve (AUC₀-₂₄h) - arm 1 vs. arm 2 | 24 hours
  Difference in plasma concentrations of yohimbine expressed as area under the curve (AUC₀-₂₄h) between women classified as CYP2D6 poor metabolizers (PM) (arm 1) and women classified as CYP2D6 extensive metabolizers (EM) (arm 2).
Yohimbine plasma concentration expressed as area under the curve (AUC₀-₂₄h) - arm 3 vs. arm 4 | 24 hours
  Difference in plasma concentrations of yohimbine expressed as area under the curve (AUC₀-₂₄h) between men classified as CYP2D6 poor metabolizers (PM) (arm 3) and men classified as CYP2D6 extensive metabolizers (EM) (arm 4).

SECONDARY OUTCOMES:
Cmax of yohimbine and 11-OH-yohimbine | 24 hours
  Differences in maximum concentration (Cmax) of yohimbine and the primary metabolite 11-OH-yohimbine between CYP2D6 poor metabolizers (PM) and extensive metabolizers (EM) within the same sex (Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4) and between women and men classified as PM (Arm 1 vs. Arm 3) and EM (Arm 2 vs. Arm 4).
tmax of yohimbine and 11-OH-yohimbine | 24 hours
  Differences in time to maximum concentration (tmax) of yohimbine and the primary metabolite 11-OH-yohimbine between CYP2D6 poor metabolizers (PM) and extensive metabolizers (EM) within the same sex (Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4) and between women and men classified as PM (Arm 1 vs. Arm 3) and EM (Arm 2 vs. Arm 4).
Clearance of yohimbine and 11-OH-yohimbine | 24 hours
  Differences in total and renal clearance of yohimbine and the primary metabolite 11-OH-yohimbine between CYP2D6 poor metabolizers (PM) and extensive metabolizers (EM) within the same sex (Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4) and between women and men classified as PM (Arm 1 vs. Arm 3) and EM (Arm 2 vs. Arm 4).
Apparent volume of distribution of yohimbine and 11-OH-yohimbine | 24 hours
  Differences in apparent volume of distribution of yohimbine and the primary metabolite 11-OH-yohimbine between CYP2D6 poor metabolizers (PM) and extensive metabolizers (EM) within the same sex (Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4) and between women and men classified as PM (Arm 1 vs. Arm 3) and EM (Arm 2 vs. Arm 4).
11-OH-Yohimbine plasma concentration expressed as area under the curve (AUC₀-₂₄h) | 24 hours
  Differences in plasma concentrations of 11-OH-yohimbine expressed as area under the curve (AUC₀-₂₄h) between CYP2D6 poor metabolizers (PM) and extensive metabolizers (EM) within the same sex (Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4) and between women and men classified as PM (Arm 1 vs. Arm 3) and EM (Arm 2 vs. Arm 4).

OTHER OUTCOMES:
Cmax of ¹³C₃-caffeine and paraxanthine | 24 hours
  Differences in maximum concentration (Cmax) of ¹³C₃-caffeine and its metabolite paraxanthine will be analyzed across all study arms and correlated with Cmax values of yohimbine and its primary metabolite 11-OH-yohimbine to assess potential interactions between CYP2D6 (involved in yohimbine metabolism) and CYP1A2 (involved in ¹³C₃-caffeine metabolism).
tmax of ¹³C₃-caffeine and paraxanthine | 24 hours
  Differences in time to maximum concentration (tmax) of ¹³C₃-caffeine and its metabolite paraxanthine will be analyzed across all study arms and correlated with tmax values of yohimbine and its primary metabolite 11-OH-yohimbine to assess potential interactions between CYP2D6 (involved in yohimbine metabolism) and CYP1A2 (involved in ¹³C₃-caffeine metabolism).
¹³C₃-caffeine and paraxanthine plasma concentrations expressed as area under the curve (AUC₀-₂₄h) | 24 hours
  Differences in plasma concentrations of ¹³C₃-caffeine and its metabolite paraxanthine expressed as area under the curve (AUC₀-₂₄h) will be analyzed across all study arms and correlated with AUC₀-₂₄h values of yohimbine and its primary metabolite 11-OH-yohimbine to assess potential interactions between CYP2D6 (involved in yohimbine metabolism) and CYP1A2 (involved in ¹³C₃-caffeine metabolism)
Renal clearance of ¹³C₃-caffeine and paraxanthine | 24 hours
  Differences in renal clearance of ¹³C₃-caffeine and its metabolite paraxanthine will be analyzed across all study arms and correlated with renal clearance values of yohimbine and its primary metabolite 11-OH-yohimbine to assess potential interactions between CYP2D6 (involved in yohimbine metabolism) and CYP1A2 (involved in ¹³C₃-caffeine metabolism).
Apparent volume of distribution of ¹³C₃-caffeine and paraxanthine | 24 hours
  Differences in apparent volume of distribution of ¹³C₃-caffeine and its metabolite paraxanthine will be analyzed across all study arms and correlated with apparent volume of distribution values of yohimbine and its primary metabolite 11-OH-yohimbine to assess potential interactions between CYP2D6 (involved in yohimbine metabolism) and CYP1A2 (involved in ¹³C₃-caffeine metabolism).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medicine Greifswald, Institute of Pharmacology, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No